CLINICAL TRIAL: NCT01132846
Title: Renal Optimization Strategies Evaluation in Acute Heart Failure and Reliable Evaluation of Dyspnea in the Heart Failure Network ROSE Study
Brief Title: Renal Optimization Strategies Evaluation in Acute Heart Failure and Reliable Evaluation of Dyspnea in the Heart Failure Network (ROSE) Study
Acronym: ROSE/RED ROSE
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Duke University (Other)
Collaborators: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: Pro00024136; U01HL084904 (NIH); Pro00029908 (Other: RED ROSE Number); Pro00023578 (Other: Duke)
Record Dates: First submitted 2010-05-27; First posted 2010-05-28 (Estimated); Results first posted 2014-08-21 (Estimated); Last update posted 2014-08-21 (Estimated); Status verified 2014-08

CONDITIONS: Acute Heart Failure
MeSH Terms: interventions — Natriuretic Peptide, Brain; Dopamine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Low dose Dopamine (Active Comparator): Drug: Dopamine
  Participants will be randomized to receive low dose dopamine or placebo during first 72 hours of participation in the study
  Interventions: Drug: Dopamine
- Placebo (Placebo Comparator): Drug: Placebo Participants will receive placebo in place of low dose dopamine or low dose nesiritide depending on randomization.
  Interventions: Other: Placebo
- Low Dose Nesiritide (Active Comparator): Participants could be randomized to receive low dose nesiritide or placebo during the first 72 hours in the trial.
  Interventions: Drug: Nesiritide

INTERVENTIONS:
Other: Placebo — Participants will be randomized to receive Low dose Dopamine or placebo plus optimal diuretic or Low dose Nesiritide or placebo plus optimal diuretic.
  Arms: Placebo
Drug: Nesiritide — Active Comparator: Low Dose Nesiritide
  Participants randomized to the low dose nesiritide arm will receive nesiritide of 0.005 ug/kg/min or placebo during the first 72 hours in the trial.
  Arms: Low Dose Nesiritide
Drug: Dopamine — Participants randomized to the low dose dopamine arm will receive dopamine of 2ug/kg/min or placebo during the first 72 hours in the trial.
  Arms: Low dose Dopamine

SUMMARY:
The purpose of this study is to determine the benefits and safety of intravenous administration of low dose nesiritide or low dose dopamine in patients with congestive heart failure and kidney dysfunction. There is a substudy in a subset of subjects that is being used to determine whether the Provocative Dyspnea Severity Score (pDSS) is a more sensitive index of variability in clinical status than the dyspnea VAS assessed without standardization of conditions at assessments.

DETAILED DESCRIPTION:
Acute heart failure (AHF) is the most common cause of hospital admission in patients over age 65, accounting for 1,000,000 admissions, over 6 million hospital days, and $12 billion in costs annually. The prognosis of patients admitted with AHF is dismal, with a 20-30% readmission rate and a 20-30% mortality rate within six months after admission. Recent studies have established the prognostic importance of renal function in patients with heart failure. In patients who are hospitalized with decompensated congestive heart failure, worsening renal function is also associated with worse outcome, Various studies have estimated that 25-30% of patients hospitalized for decompensated CHF have worsening of renal function leading to prolonged hospitalization, increased morbidity and mortality. Although there are no FDA approved renal adjuvant therapies for AHF, several novel adjuvant therapies for use in AHF are being investigated in randomized clinical trials. Additionally, there are currently available strategies, with the potential for improving renal function in AHF such as low dose dopamine and low dose nesiritide. However, these strategies have not been investigated.

Participation in this study will last 6 months. All potential participants will undergo initial screening, which wil include a medical history, physical exam, blood draws, measurements of fluid intake and output, and questionnaires. The same evaluations and procedures will be repeated at various points during the study. Eligible participants will be randomly assigned to receive low dose nesiritide or placebo with optimal diuretic dosing or low dose dopamine or placebo with optimal diuretic dosing.

Follow-up assessments will occur at Baseline, 24 hours, 48 hours, 72 hours, day 7 or discharge, day 60 and 6 months. Follow-up assessments will include medical history, physical exam, blood draws, measurements of fluid intake and output, questionnaires and questions about medications and changes in health.

The RED ROSE substudy involves a subset of ROSE patients in looking at the dyspnea assessment. The dyspnea visual analog scale (dyspnea VAS) has been suggested to be superior to other ordinal (Likert) scales in assessment of dyspnea in acute heart failure syndromes (AHFS)1. However, there is no standardization of conditions (oxygen supplementation, position, activity) at the time of VAS assessment and thus, it may not optimally reflect the variability in dyspnea severity in AHFS patients. This insensitivity to variability at baseline and subsequent assessment may limit the ability to reflect variation in response over time and with alternate treatment strategies. A standardized and sequentially provocative assessment of dyspnea (provocative dyspnea severity score, pDSS) may better reflect variation in dyspnea severity and variation in response over time and with alternate treatment strategies. Substudy subjects will be asked to complete a provocative dyspnea assessment at baseline, 24, 48 and 72 hours. The subjects will be asked to complete a 6 minute walk assessment at the 72 hour visit.

ELIGIBILITY:
Inclusion Criteria:

* A diagnosis of heart failure as defined by the presence of at least 1 symptom (dyspnea, orthopnea, or edema) AND 1 sign (rales on auscultation, peripheral edema, ascites, pulmonary vascular congestion on chest radiography)
* Prior clinical diagnosis of heart failure Must be identified within 24 hours of hospital admission (24 hour clock begins when the admission orders are placed)
* Estimated GFR of > 15 but < 60 mL/min/1.73m2 determined by the MDRD equation
* Male or female patient ≥18 years old
* Willingness to provide informed consent
* Ability to have a PICC or central line placed (if needed) within 12 hours of randomization and study drug infusion started
* Anticipated hospitalization of at least 72 hours

Exclusion Criteria:

* Received IV vasoactive treatment or ultra-filtration therapy for heart failure since initial presentation
* Anticipated need for IV vasoactive treatment or ultra-filtration for heart failure during this hospitalization
* Systolic BP <90 mmHg
* Hemoglobin (Hgb) < 9 g/dl
* Renal replacement therapy
* History of renal artery stenosis > 50%
* Hemodynamically significant arrhythmias including ventricular tachycardia or defibrillator shock within 4 weeks
* Acute coronary syndrome within 4 weeks as defined by electrocardiographic (ECG) ST-segment depression or prominent T-wave inversion and/or positive biomarkers of necrosis (e.g., troponin) in the absence of ST-segment elevation and in an appropriate clinical setting (chest discomfort or anginal equivalent)
* Active myocarditis
* Hypertrophic obstructive cardiomyopathy
* Greater than moderate stenotic valvular disease
* Restrictive or constrictive cardiomyopathy
* Complex congenital heart disease
* Constrictive pericarditis
* Non-cardiac pulmonary edema
* Clinical evidence of digoxin toxicity
* Need for mechanical hemodynamic support
* Sepsis
* Terminal illness (other than HF) with expected survival of less than 1 year
* Previous adverse reaction to the study drugs
* Use of IV iodinated radiocontrast material in last 72 hours or planned during hospitalization
* Enrollment or planned enrollment in another randomized clinical trial during this hospitalization
* Inability to comply with planned study procedures
* Pregnancy or nursing mothers

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 360 (Actual)
Dates: Start 2010-08; Primary Completion 2013-05 (Actual); Study Completion 2013-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Kerry L Lee, PhD, Principal Investigator — Duke University; Eugene Braunwald, MD, Study Chair — Harvard University
Locations (8):
- United States (7):
  - Brigham and Women's Hospital, Boston, Massachusetts
  - Minnesota Heart Failure Network, Minneapolis, Minnesota
  - Mayo Clinic, Rochester, Minnesota
  - Duke University Medical Center, Durham, North Carolina
  - Baylor College of Medicine, Houston, Texas
  - University of Utah Health Sciences Center, Murry, Utah
  - University of Vermont- Fletcher Allen Health Care, Burlington, Vermont
- Montreal Heart Institute, Montreal, Quebec, Canada

REFERENCES:
- [Result] Chen HH, Anstrom KJ, Givertz MM, Stevenson LW, Semigran MJ, Goldsmith SR, Bart BA, Bull DA, Stehlik J, LeWinter MM, Konstam MA, Huggins GS, Rouleau JL, O'Meara E, Tang WH, Starling RC, Butler J, Deswal A, Felker GM, O'Connor CM, Bonita RE, Margulies KB, Cappola TP, Ofili EO, Mann DL, Davila-Roman VG, McNulty SE, Borlaug BA, Velazquez EJ, Lee KL, Shah MR, Hernandez AF, Braunwald E, Redfield MM; NHLBI Heart Failure Clinical Research Network. Low-dose dopamine or low-dose nesiritide in acute heart failure with renal dysfunction: the ROSE acute heart failure randomized trial. JAMA. 2013 Dec 18;310(23):2533-43. doi: 10.1001/jama.2013.282190. PMID 24247300
- [Derived] Adel FW, Rikhi A, Wan SH, Iyer SR, Chakraborty H, McNulty S, Tang WHW, Felker GM, Givertz MM, Chen HH. Annexin A1 is a Potential Novel Biomarker of Congestion in Acute Heart Failure. J Card Fail. 2020 Aug;26(8):727-732. doi: 10.1016/j.cardfail.2020.05.012. Epub 2020 May 27. PMID 32473378
- [Derived] Kelly JP, Cooper LB, Gallup D, Anstrom KJ, Chen HH, Redfield MM, O'Connor CM, Mentz RJ, Hernanadez AF, Felker GM. Implications of Using Different Definitions on Outcomes in Worsening Heart Failure. Circ Heart Fail. 2016 Aug;9(8):e003048. doi: 10.1161/CIRCHEARTFAILURE.116.003048. PMID 27514750
- [Derived] Wan SH, Stevens SR, Borlaug BA, Anstrom KJ, Deswal A, Felker GM, Givertz MM, Bart BA, Tang WH, Redfield MM, Chen HH. Differential Response to Low-Dose Dopamine or Low-Dose Nesiritide in Acute Heart Failure With Reduced or Preserved Ejection Fraction: Results From the ROSE AHF Trial (Renal Optimization Strategies Evaluation in Acute Heart Failure). Circ Heart Fail. 2016 Aug;9(8):10.1161/CIRCHEARTFAILURE.115.002593 e002593. doi: 10.1161/CIRCHEARTFAILURE.115.002593. PMID 27512103
- [Derived] de Denus S, Rouleau JL, Mann DL, Huggins GS, Cappola TP, Shah SH, Keleti J, Zada YF, Provost S, Bardhadi A, Phillips MS, Normand V, Mongrain I, Dube MP. A pharmacogenetic investigation of intravenous furosemide in decompensated heart failure: a meta-analysis of three clinical trials. Pharmacogenomics J. 2017 Mar;17(2):192-200. doi: 10.1038/tpj.2016.4. Epub 2016 Mar 1. PMID 26927285
- [Derived] Chen HH, AbouEzzeddine OF, Anstrom KJ, Givertz MM, Bart BA, Felker GM, Hernandez AF, Lee KL, Braunwald E, Redfield MM; Heart Failure Clinical Research Network. Targeting the kidney in acute heart failure: can old drugs provide new benefit? Renal Optimization Strategies Evaluation in Acute Heart Failure (ROSE AHF) trial. Circ Heart Fail. 2013 Sep 1;6(5):1087-94. doi: 10.1161/CIRCHEARTFAILURE.113.000347. No abstract available. PMID 24046475

RESULTS

PARTICIPANT FLOW:
Groups:
- Low Dose Dopamine: Drug: Dopamine
  Participants will be randomized to receive low dose dopamine or placebo during first 72 hours of participation in the study
  Dopamine: Participants randomized to the low dose dopamine arm will receive dopamine of 2ug/kg/min or placebo during the first 72 hours in the trial.
- Placebo: Drug: Placebo
  Participants will receive placebo in place of low dose dopamine or low dose nesiritide depending on randomization.
  Placebo: Participants will be randomized to receive Low dose Dopamine or placebo plus optimal diuretic or Low dose Nesiritide or placebo plus optimal diuretic.
- Low Dose Nesiritide: Drug: Nesiritide
  Participants could be randomized to receive low dose nesiritide or placebo during the first 72 hours in the trial.
  Participants randomized to the low dose nesiritide arm will receive nesiritide of 0.005 ug/kg/min or placebo during the first 72 hours in the trial.
Period: Overall Study
Arm/Group | Low Dose Dopamine | Placebo | Low Dose Nesiritide
Started | 122 | 119 | 119
Completed | 106 | 101 | 108
Not Completed | 16 | 18 | 11

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Low Dose Dopamine | Placebo | Low Dose Nesiritide | Total
Number analyzed (Participants) | 122 | 119 | 119 | 360
Age, Continuous [Mean (Standard Deviation); unit: years] | 71.0 (11.1) | 69.3 (12.6) | 68.3 (13.0) | 69.6 (12.3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 38 | 30 | 28 | 96
  Male | 84 | 89 | 91 | 264
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 3 | 1 | 3 | 7
  Asian | 1 | 1 | 1 | 3
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 27 | 23 | 24 | 74
  White | 90 | 91 | 91 | 272
  More than one race | 1 | 1 | 0 | 2
  Unknown or Not Reported | 0 | 2 | 0 | 2
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 6 | 5 | 3 | 14
  Not Hispanic or Latino | 116 | 112 | 116 | 344
  Unknown or Not Reported | 0 | 2 | 0 | 2

OUTCOME MEASURES:

1. Primary Outcome: Change in Cystatin C
Description: The primary Safety endpoint is change in serum cystatin C from randomization to 72 hours.
Time Frame: Randomization to 72 hours
Measure: Mean (Standard Deviation); unit: mg/L
Arm/Group | Low Dose Dopamine | Placebo | Low Dose Nesiritide
Number analyzed (Participants) | 122 | 119 | 119
mg/L | .12 (.32) | .11 (.27) | .07 (.34)

2. Primary Outcome: Change in Dyspnea Assessment (RED-ROSE Substudy)
Description: To determine whether the pDSS is a more sensitive index of variability in dyspnea status than the dyspnea VAS assessed without standardization of conditions at assessment as assessed by change in Dyspnea VAS.
  Dyspnea VAS range -100 to + 100 Larger number is better
Time Frame: Baseline to 72 hours
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Low Dose Dopamine | Placebo | Low Dose Nesiritide
Number analyzed (Participants) | 70 | 70 | 73
units on a scale | 16.1 (30.7) | 16.2 (22.3) | 16.8 (24.2)

3. Primary Outcome: Decongestive Changes- RED-ROSE
Description: To determine whether changes in pDSS or dyspnea VAS are related to the response to decongestive therapy as evidenced by fluid volume loss
  Fluid volume loss is defined as cumulative urinary output minus fluid intake during the first 72 hours post randomization.
Time Frame: Baseline to 72 hours
Population: RED-ROSE is a substudy of the overall ROSE study. Only consented and enrolled RED-ROSE subjects participated.
Measure: Mean (Standard Deviation); unit: mL
Arm/Group | Low Dose Dopamine | Placebo | Low Dose Nesiritide
Number analyzed (Participants) | 74 | 72 | 72
mL | 4526.0 (3191.9) | 4659.9 (2862.5) | 5177.2 (2830.5)

4. Primary Outcome: Cumulative Urinary Volume
Description: The primary efficacy endpoint is cumulative urinary volume (UV; +/- indwelling urinary catheter) at 72 hours
Time Frame: Randomization to 72 hours
Measure: Mean (Standard Deviation); unit: mL
Arm/Group | Low Dose Dopamine | Placebo | Low Dose Nesiritide
Number analyzed (Participants) | 122 | 119 | 119
mL | 8524 (3418) | 8296 (2973) | 8574 (3115)

5. Secondary Outcome: Change in Weight
Description: Change in weight from randomization to 72 hours. Secondary Endpoint
Time Frame: randomization to 72 hours
Measure: Mean (Standard Deviation); unit: lbs
Arm/Group | Low Dose Dopamine | Placebo | Low Dose Nesiritide
Number analyzed (Participants) | 122 | 119 | 119
lbs | -7.40 (7.94) | -7.73 (7.04) | -7.15 (7.80)

6. Secondary Outcome: Worst Reported Symptom Changes-RED-ROSE
Description: To determine whether changes in worst reported symptom (WRS) (dyspnea, body swelling or fatigue) VAS (WRS-VAS) are related to the response to decongestive therapy as assessed by change in WRS VAS.
  WRS range -100 to + 100 Higher number is better (improved)
Time Frame: Change from Baseline to 72 hours
Population: RED-ROSE was a substudy of the main ROSE study. Only subjects consented and enrolled in RED-ROSE were included in this analysis.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Low Dose Dopamine | Placebo | Low Dose Nesiritide
Number analyzed (Participants) | 68 | 70 | 73
units on a scale | 20.9 (29.6) | 19.6 (22.7) | 25.6 (25.6)

7. Secondary Outcome: Change in Clinical Stability- RED-ROSE
Description: Change in clinical stability as assessed by 60 day death, re-hospitalization or unscheduled outpatient visit
Time Frame: Baseline to 60 days
Population: RED-ROSE was a substudy of the main ROSE trial. Only subjects consented and enrolled in RED-ROSE were included in this analysis.
Measure: Number; unit: participants
Arm/Group | Low Dose Dopamine | Placebo | Low Dose Nesiritide
Number analyzed (Participants) | 76 | 75 | 76
participants | 30 | 34 | 27

8. Secondary Outcome: Change in Serum Creatinine
Time Frame: randomization to 72 hours
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | Low Dose Dopamine | Placebo | Low Dose Nesiritide
Number analyzed (Participants) | 122 | 119 | 119
mg/dL | 0.00 (0.44) | 0.02 (0.33) | 0.02 (0.42)

9. Secondary Outcome: Dyspnea Visual Analog Scale Area Under the Curve
Description: Range 0 to 7200 Higher is better
Time Frame: randomization to 72 hours
Population: Based upon data completeness, sample size for this endpoint does not match the overall ROSE population.
Measure: Mean (Standard Deviation); unit: units on a scale * hours
Arm/Group | Low Dose Dopamine | Placebo | Low Dose Nesiritide
Number analyzed (Participants) | 112 | 114 | 115
units on a scale * hours | 4935.8 (1472.1) | 4997.6 (1479.9) | 4831.4 (1294.1)

10. Secondary Outcome: Change in Heart Failure Status
Description: Persistent or worsening heart failure defined as need for rescue therapy.
Time Frame: randomization to 72 hours
Population: Based upon data completeness, sample size for this endpoint does not match the overall ROSE population.
Measure: Number; unit: participants
Arm/Group | Low Dose Dopamine | Placebo | Low Dose Nesiritide
Number analyzed (Participants) | 118 | 116 | 117
participants | 11 | 5 | 6

11. Secondary Outcome: Change in Treatment Response
Description: Treatment failure including any of the following:
  * development of cardio-renal syndrome
  * worsening/persistent heart failure
  * significant hypotension requiring discontinuation of study drug
  * significant tachycardia requiring discontinuation of study drug death
Time Frame: randomization to 72 hours
Population: Based upon data completeness, sample size for this endpoint does not match the overall ROSE population.
Measure: Number; unit: participants
Arm/Group | Low Dose Dopamine | Placebo | Low Dose Nesiritide
Number analyzed (Participants) | 117 | 115 | 119
participants | 35 | 32 | 48

12. Secondary Outcome: Cumulative Urinary Sodium Excretion
Time Frame: Randomization to 72 hours
Measure: Mean (Standard Deviation); unit: mmol
Arm/Group | Low Dose Dopamine | Placebo | Low Dose Nesiritide
Number analyzed (Participants) | 122 | 119 | 119
mmol | 527.0 (299.0) | 539.8 (302.7) | 515.2 (261.4)

13. Secondary Outcome: Change in Blood Urea Nitrogen (BUN)/ Serum Cystatin C Ratio
Description: BUN measured in mg/dL Cystatin C measured in mg/L
  No units were used in calculated the ratio
Time Frame: Randomization to 72 hours
Measure: Mean (Standard Deviation); unit: ratio
Arm/Group | Low Dose Dopamine | Placebo | Low Dose Nesiritide
Number analyzed (Participants) | 122 | 119 | 119
ratio | -2.34 (25.33) | 0.23 (5.16) | 0.74 (7.60)

14. Secondary Outcome: Development of Cardio-renal Syndrome
Time Frame: Randomization to 72 hours
Population: Based upon data completeness, sample size for this endpoint does not match the overall ROSE population.
Measure: Number; unit: participants
Arm/Group | Low Dose Dopamine | Placebo | Low Dose Nesiritide
Number analyzed (Participants) | 105 | 110 | 111
participants | 23 | 24 | 28

15. Secondary Outcome: Global Visual Analog Scale Area Under the Curve
Description: Range 0 to 7200 Higher is better/improved
Time Frame: Randomization to 72 hours
Population: Based upon data completeness, sample size for this endpoint does not match the overall ROSE population.
Measure: Mean (Standard Deviation); unit: units on a scale * hours
Arm/Group | Low Dose Dopamine | Placebo | Low Dose Nesiritide
Number analyzed (Participants) | 112 | 113 | 114
units on a scale * hours | 4553.4 (1324.9) | 4703.6 (1403.4) | 4498.3 (1301.5)

ADVERSE EVENTS:
Arm/Group | Low Dose Dopamine | Placebo | Low Dose Nesiritide
Serious Adverse Events (participants affected / at risk) | 30/122 | 24/119 | 21/119
Other Adverse Events (participants affected / at risk) | 0/122 | 0/119 | 0/119
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Low Dose Dopamine (N=122) | Placebo (N=119) | Low Dose Nesiritide (N=119)
Anemia (Blood and lymphatic system disorders) | 1 | 2 | 0
Hemorrhagic Anemia (Blood and lymphatic system disorders) | 1 | 0 | 0
Acute Myocardial Infarction (Cardiac disorders) | 1 | 0 | 0
Atrioventricular Block, Second Degree (Cardiac disorders) | 1 | 0 | 0
Cardiac Arrest (Cardiac disorders) | 2 | 2 | 0
Paroxysmal Arrhythmia (Cardiac disorders) | 0 | 1 | 0
Ventricular Arrhythmia (Cardiac disorders) | 0 | 2 | 0
Ear Pain (Ear and labyrinth disorders) | 0 | 0 | 1
Visual Impairment (Eye disorders) | 0 | 0 | 1
Abdominal Pain (Gastrointestinal disorders) | 0 | 0 | 1
Constipation (Gastrointestinal disorders) | 0 | 0 | 1
Diarrhea (Gastrointestinal disorders) | 1 | 1 | 0
Gastroesophogeal Reflux Disease (Gastrointestinal disorders) | 1 | 0 | 0
Lower Gastrointestinal Hemorrhage (Gastrointestinal disorders) | 1 | 2 | 1
Melaena (Gastrointestinal disorders) | 0 | 0 | 1
Upper Gastrointestinal Hemorrhage (Gastrointestinal disorders) | 0 | 0 | 1
Vomitting (Gastrointestinal disorders) | 1 | 0 | 0
Infusion Site Irritation (General disorders) | 1 | 0 | 0
Chest Discomfort (General disorders) | 0 | 0 | 1
Chest Pain (General disorders) | 0 | 0 | 1
Death (General disorders) | 0 | 0 | 1
Cellulitis (Infections and infestations) | 1 | 0 | 0
Influenza (Infections and infestations) | 2 | 0 | 0
Osteomyelitis (Infections and infestations) | 0 | 1 | 0
Pneumonia (Infections and infestations) | 2 | 1 | 1
Sepsis (Infections and infestations) | 4 | 2 | 0
Septic Shock (Infections and infestations) | 1 | 0 | 0
Upper Respiratory Tract Infections (Infections and infestations) | 1 | 0 | 0
Fall (Injury, poisoning and procedural complications) | 0 | 1 | 0
Procedural Complications (Injury, poisoning and procedural complications) | 1 | 0 | 0
Anticoagulation Drug Level Above Therapeutic (Investigations) | 2 | 0 | 0
Weight Decreased (Investigations) | 0 | 1 | 0
Hypoglycemia (Metabolism and nutrition disorders) | 2 | 1 | 1
Hyperammonaemia (Metabolism and nutrition disorders) | 0 | 0 | 1
Cerebrovascular Accident (Nervous system disorders) | 1 | 1 | 1
Syncope (Nervous system disorders) | 0 | 2 | 2
Basal Cell Carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1
Renal Failure (Renal and urinary disorders) | 0 | 3 | 0
Acute Respiratory Failure (Respiratory, thoracic and mediastinal disorders) | 2 | 0 | 0
Respiratory Failure (Respiratory, thoracic and mediastinal disorders) | 2 | 1 | 0
Hypotension (Vascular disorders) | 2 | 7 | 5

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No